CLINICAL TRIAL: NCT07020442
Title: Department of Sport Performance, National Taiwan University of Sport
Brief Title: Effects of Integrated Neuromuscular Training on Physical Fitness in Badminton Athletes With Different Maturity Statuses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research has been completed
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chen Che Hsiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHChen
Record Dates: First submitted 2025-04-10; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Athletic Injuries
Keywords: strength; asymmetry; maturation; injury
MeSH Terms: conditions — Athletic Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: 24 well-trained male badminton players (age: 13.5 ± 1.15 years), grouped by maturation status (pre- and post-peak height velocity; n = 12 each). All participants completed two NMT sessions weekly. Pre- and post-training assessments included 20-m sprint, countermovement jump (CMJ), agility T-test, hexagon test, and Y-balance test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (pre maturation status (Experimental): maturation status (pre peak height velocity; n = 12 each).
  Interventions: Other: integrated neuromuscular training
- post maturation status (Experimental): maturation status (post peak height velocity; n = 12 each).
  Interventions: Other: integrated neuromuscular training

INTERVENTIONS:
Other: integrated neuromuscular training — a 12-week integrated neuromuscular training (NMT) program. All participants completed two NMT sessions weekly.

SUMMARY:
Dominant leg use in badminton may contribute to lower limb asymmetry, potentially affecting performance and injury risk. This study investigated the effects of a 12-week integrated neuromuscular training (NMT) program on sport performance in 24 well-trained male badminton players, grouped by maturation status (pre- and post-peak height velocity; n = 12 each). All participants completed two NMT sessions weekly. Pre- and post-training assessments included 20-m sprint, countermovement jump (CMJ), agility T-test, hexagon test, and Y-balance test.

DETAILED DESCRIPTION:
This study aimed to evaluate the effects of integrated NMT on lower extremity sports performance in pre-PHV and post-PHV male badminton players. A parallel, two-group, stratified randomized controlled design was employed. The intervention lasted 12 weeks, with two sessions per week. All dependent variables were assessed at baseline and after 12 weeks. Following the training period, participants completed sport-specific performance tests, including the 20-m linear sprint, countermovement jump, agility T-test, hexagon test, and Y-balance test.Twenty-four well-trained male badminton players with a mean age of 13.5 ± 1.15 years participated in this study . The results of this study underscore the importance of maturation status in determining how youth athletes respond to integrated NMT interventions.

ELIGIBILITY:
Inclusion Criteria:

- Male badminton athletes with no lower limb injuries within 6 months

Exclusion Criteria:

* Female athletes and athletes with lower limb injuries

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
20-m linear sprint test | Baseline and immediately after the intervention
  A 20-m linear sprint test was conducted using a Smartspeed Pro timing gate system
Countermovement jump | Baseline and immediately after the intervention
  The participants stood on a jump mat (Smart Jump, Fusion Sport, Brisbane, Australia) with both hands placed on hips, and participants were instructed to perform a countermovement
Agility T-Test | Baseline and immediately after the intervention
  The agility T-test was conducted using a Smartspeed Pro timing gate system
Hexagon test | Baseline and immediately after the intervention
  The test has been used measure of agility and food quickness. The test began with the participants standing on the tape strip placed in the middle of the hexagon, facing forward in the middle of a hexagon measuring 60 cm per side and with each angle being120-degree.
Y-balance test | Baseline and immediately after the intervention
  The test involved unilateral lower limb reaches in three directions: anterior (A), postero-medial (PM), and postero-lateral (PL). Participants completed three official trials in each direction. During each trial, participants kept their hands on their hips while reaching with the non-stance leg while barefoot, ensuring that the stance heel remained in contact with the ground.

CONTACTS AND LOCATIONS:
Overall Officials: CHEN CHE HSIU, Professor, Principal Investigator — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No